CLINICAL TRIAL: NCT05353985
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study to Evaluate the Efficacy and Safety of TAK-062 for the Treatment of Active Celiac Disease in Subjects Attempting a Gluten-Free Diet
Brief Title: A Study of TAK-062 in Treatment of Active Celiac Disease in Participants Attempting a Gluten-Free Diet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-062-2001; 2020-005438-14 (EudraCT Number)
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Celiac Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: TAK-062 Placebo + SIGE Gluten-Bar (Placebo Comparator): TAK-062 placebo-matching 4 tablets, orally, taken within pre-determined time before the start of a meal and SIGE gluten bar, orally, with a meal, at protocol defined timepoints, for up to 24 weeks.
  Interventions: Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-Bar; Drug: TAK-062 Placebo
- Cohort 1: TAK-062 Dose 1 + SIGE Gluten-Bar (Experimental): TAK-062 Dose 1, 4 tablets, orally, taken within pre-determined time before the start of a meal and SIGE gluten bar, orally, with a meal, at protocol defined timepoints, for up to 24 weeks.
  Interventions: Drug: TAK-062; Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-Bar
- Cohort 2: TAK-062 Placebo + SIGE Gluten-Bar (Placebo Comparator): TAK-062 placebo-matching 4 tablets, orally, taken within pre-determined time before the start of a meal and SIGE gluten bar, orally, with a meal, at protocol defined timepoints, for up to 24 weeks.
  Interventions: Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-Bar; Drug: TAK-062 Placebo
- Cohort 2: TAK-062 Dose 2 + SIGE Gluten-Bar (Experimental): TAK-062 Dose 2, 4 tablets, orally, taken within pre-determined time before the start of a meal and SIGE gluten bar, orally, with a meal, at protocol defined timepoints, for up to 24 weeks.
  Interventions: Drug: TAK-062; Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-Bar
- Cohort 2: TAK-062 Dose 3 + SIGE Gluten-Bar (Experimental): TAK-062 Dose 3, 4 tablets, orally, taken within pre-determined time before the start of a meal and SIGE gluten bar, orally, with a meal, at protocol defined timepoints, for up to 24 weeks.
  Interventions: Drug: TAK-062; Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-Bar
- Cohort 2: TAK-062 Placebo + Gluten-free SIGE Bar (Placebo Comparator): TAK-062 placebo-matching 4 tablets, orally, taken within pre-determined time before the start of a meal and gluten-free SIGE bar, orally, with a meal, at protocol defined timepoints, for up to 24 weeks.
  Interventions: Drug: TAK-062 Placebo; Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-free Bar
- Cohort 2: TAK-062 Dose 1 + Gluten-free SIGE Bar (Experimental): TAK-062 Dose 1, 4 tablets, orally, taken within pre-determined time before the start of a meal and gluten-free SIGE bar, orally, with a meal, at protocol defined timepoints, for up to 24 weeks.
  Interventions: Drug: TAK-062; Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-free Bar
- Cohort 2: TAK-062 Dose 2 + Gluten-free SIGE Bar (Experimental): TAK-062 4 tablets, orally, taken within pre-determined time before the start of a meal and gluten-free SIGE bar, orally, with a meal, at protocol defined timepoints, for up to 24 weeks.
  Interventions: Drug: TAK-062; Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-free Bar

INTERVENTIONS:
Drug: TAK-062 — TAK-062 tablets.
  Arms: Cohort 1: TAK-062 Dose 1 + SIGE Gluten-Bar; Cohort 2: TAK-062 Dose 1 + Gluten-free SIGE Bar; Cohort 2: TAK-062 Dose 2 + Gluten-free SIGE Bar; Cohort 2: TAK-062 Dose 2 + SIGE Gluten-Bar; Cohort 2: TAK-062 Dose 3 + SIGE Gluten-Bar
Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-Bar — SIGE gluten bars.
  Arms: Cohort 1: TAK-062 Dose 1 + SIGE Gluten-Bar; Cohort 1: TAK-062 Placebo + SIGE Gluten-Bar; Cohort 2: TAK-062 Dose 2 + SIGE Gluten-Bar; Cohort 2: TAK-062 Dose 3 + SIGE Gluten-Bar; Cohort 2: TAK-062 Placebo + SIGE Gluten-Bar
Drug: TAK-062 Placebo — TAK-062 placebo-matching tablets.
  Arms: Cohort 1: TAK-062 Placebo + SIGE Gluten-Bar; Cohort 2: TAK-062 Placebo + Gluten-free SIGE Bar; Cohort 2: TAK-062 Placebo + SIGE Gluten-Bar
Dietary Supplement: Simulated Inadvertent Gluten Exposure (SIGE) Gluten-free Bar — SIGE gluten-free bars.
  Arms: Cohort 2: TAK-062 Dose 1 + Gluten-free SIGE Bar; Cohort 2: TAK-062 Dose 2 + Gluten-free SIGE Bar; Cohort 2: TAK-062 Placebo + Gluten-free SIGE Bar

SUMMARY:
The main aim is to see how TAK-062 works to reduce celiac-related symptoms and improve small intestinal damage due to gluten exposure, in participants with celiac disease (CeD) attempting to maintain a gluten-free diet (GFD) in treated participants versus placebo controls.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-062. TAK-062 is designed to break down gluten in the stomach and is being tested to treat people who have active CeD, attempting to maintain a GFD.

The study will enroll approximately 357 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups in Cohort 1:

1. Cohort 1 (Age 18 and older): TAK-062 Placebo + SIGE Gluten-Bar
2. Cohort 1 (Age 18 and older): TAK-062 Dose 1 + SIGE Gluten-Bar

After the interim analysis (IA), Cohort 1 data will be reviewed by an external independent data monitoring committee (DMC), and based on the Sponsor's decision, adolescent participants will be enrolled in Cohort 2. Adult participants, 18 years and older will be enrolled into Cohort 2 once Cohort 1 has completed enrolment. Adult participants will be randomly assigned to one of the five study drug and SIGE treatment groups (Groups a-e), and approximately 21 adolescent participants will be enrolled and randomly assigned to Groups d, e, and f (adolescents only). Adolescents in Cohort 2 will receive only gluten-free SIGE bars.

1. Cohort 2 (Age 18 and older): TAK-062 Placebo + SIGE Gluten-Bar
2. Cohort 2 (Age 18 and older): TAK-062 Dose 2 + SIGE Gluten-Bar
3. Cohort 2 (Age 18 and older): TAK-062 Dose 3 + SIGE Gluten-Bar
4. Cohort 2 (Age 12 and older): TAK-062 Placebo + Gluten-free SIGE Bar
5. Cohort 2 (Age 12 and older): TAK-062 Dose 1 + Gluten-free SIGE Bar
6. Cohort 2 (Age 12-17): TAK-062 Dose 2 + Gluten-free SIGE Bar

This multi-center trial will be conducted in the United States (US), Canada, United Kingdom and the European Union. The overall time to participate in this study is approximately 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Has an adequate comprehension of a gluten-free diet (GFD) assessed by the site investigator after review of responses to a knowledge test. The final determination of a participant's adequate comprehension of a GFD is at the discretion of the investigator.
2. Has at least 1 CeD-related GI symptom of moderate or greater severity, as measured by the CDSD, on at least 3 days out of any consecutive 7-day period during the screening period (Week -8 visit until Week -4 visit), felt by the investigator to be related to gluten exposure. The CeD-related symptom(s) may vary day by day as long as the severity of at least 1 symptom is moderate or greater. The participants must meet symptom criteria to undergo esophagogastroduodenoscopy (EGD)/video capsule endoscopy (VCE).
3. Has been attempting to maintain a GFD for at least 12 months as self-reported by the participant.
4. Has small intestinal villous atrophy on duodenal biopsy defined as Vh:Cd <2.5 at Week -4.
5. The participant is human leukocyte antigen (HLA)-DQ2 and/or HLA-DQ8 positive.
6. The participant is in a good general state of health according to clinical history and physical examination, in the opinion of the investigator.
7. Have a body mass index (BMI) between 16 and 45 kilogram per meter square (kg/m^2), inclusive.

   Note: Individuals with BMI of 40 to 45 should be discussed with the medical monitor and confirmed to be appropriate for endoscopy according to local site guidelines.
8. The participant is willing and able to continue any current dietary and/or medical regimens (including gastric acid suppression) in effect at the first visit (Visit 1).

There should be no changes to diet, medications (prescription or over-the-counter) or supplements during study participation.

Exclusion Criteria:

1. Has the presence of other inflammatory GI disorders or systemic autoimmune diseases that either have the potential to cause persistent GI symptoms similar to CeD or are not well controlled without the use of excluded medication.

   * Examples of conditions that are exclusionary include inflammatory bowel disease, eosinophilic esophagitis, gastroenteritis or colitis, microscopic colitis diagnosed at screening or requiring treatment in the 6 months before screening.
   * Examples of conditions that may be permissible after discussion with the medical monitor include systemic autoimmune disease such as scleroderma, psoriatic or rheumatoid arthritis, or lupus that is stable and without GI involvement; well controlled autoimmune thyroid disease; well-controlled type 1 diabetes; or proton pump inhibitor (PPI) responsive eosinophilic esophagitis in symptomatic and histologically confirmed remission.
2. Has ongoing systemic immunosuppressant, systemic corticosteroid treatment excluding medication given for the endoscopies, or treatment with systemic immunosuppressants or systemic corticosteroids in the 12 weeks before Screening.

   • The participant is receiving immunosuppressive doses of corticosteroids: 3 mg per day or more of budesonide for more than 3 consecutive days within 3 months before Screening, more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more within 90 days before the first dose, any dose of oral or intravenous (IV) corticosteroids within 30 days of the first dose, or high-dose inhaled corticosteroids (>960 micrograms per day [μg/day] of beclomethasone dipropionate or equivalent), or other systemic immunosuppressive agents.
3. Has ongoing use of over-the-counter digestive enzymes or digestive supplements, other than lactase, including those for gluten digestion. Probiotics are allowable if they were started before Screening and not discontinued or changed in dose or type during the study.
4. Has completed the CDSD on ≤75% of the evaluable days during the run-in period until randomization.
5. Has active microscopic colitis requiring treatment in the 6 months before Screening.

   • Microscopic colitis detected at screening if sigmoidoscopy is performed would exclude the participant.
6. Has known or suspected type 2 refractory CeD or ulcerative jejunitis.
7. Has ongoing chronic use (defined as >7 days continuous use) of a nonsteroidal anti-inflammatory drug aside from <100 mg aspirin, daily, for prophylactic use.
8. Has ongoing use, or use in the 3 months before screening, of medications known to cause villous abnormalities (e.g., mycophenolate mofetil, angiotensin receptor blockers, colchicine).
9. Has used treatments for GI symptoms including antiemetics, antidiarrheals, antispasmodics, medical marijuana, (use of medical marijuana indicated for non-GI conditions is not exclusionary) within 2 weeks of Screening and during the run-in period. Participants on stable dose (i.e., more than 4 weeks) of an osmotic, bulking-forming or emollient (surface active agent) laxative are eligible, provided symptoms are considered not related to CeD in the opinion of the investigator.
10. Has a known or suspected severe enteric infection (viral, bacterial, or parasitic) within 6 months before randomization. Severe enteric infection is defined as requiring emergency room visit or hospitalization or treatment with antibiotics or anti-infectives due to infection. Non enteric viral infections, either resolved or well-controlled are not exclusionary.
11. Has a contraindication to endoscopy with duodenal biopsy.

    --Contraindication to VCE (strictures, anastomoses, etc) is not an exclusion if the participant is able to complete the other aspects of the study.
12. Has additional food allergies (tapioca syrup, oats, almonds, rice crisp, chocolate, almond, butter, wheat gluten, cocoa butter, oat flour, glycerin, sunflower lecithin, salt, and natural flavors) to nongluten ingredients in the SIGE bar study food or significant symptoms upon ingestion of the gluten-free SIGE bar during screening.
13. Has a history of intolerance, hypersensitivity, or idiosyncratic reaction to an aminoglycoside.
14. Has a known human immunodeficiency virus (HIV) infection or positive tests for hepatitis B or C. The participant has a known clinically significant chronically active hepatopathy of any origin, including cirrhosis, and participants with persistent positive hepatitis B virus surface antigen and quantitative hepatitis B virus polymerase chain reaction (PCR), or positive serology for hepatitis C virus (HCV) and quantitative HCV PCR within 6 months before the screening visit.
15. Is positive for severe acute respiratory syndrome coronavirus 2 at the time of screening and exhibits symptoms that, in the opinion of the investigator, may interfere with study compliance, completion, or accurate assessment of study outcomes or safety.
16. Has a known hypersensitivity reaction and/or allergy, including anaphylaxis, to wheat and/or gluten.
17. Has known history of hypersensitivity, idiosyncratic reaction, or intolerance to any ingredients or excipients in TAK-062 and/or placebo.
18. The participant has a current diagnosis of active malignancy or is receiving treatment for active malignancy (hormone therapy alone is not exclusionary). Participants with fully resected Stage 0 (carcinoma in situ) or Stage 1 tumor without signs of recurrence may participate. All other individuals with malignancies diagnosed in the 5 years prior to screening are excluded.

Region-specific Exclusion Criteria:

18. Participant enrolling in a study in France is not affiliated to a social security scheme or a beneficiary of such a scheme.

19. Participant enrolling in a study in France is deprived of their liberty by a judicial or administrative decision.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (102):
- United States (61):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Research Solutions of Arizona, PC, Litchfield Park, Arizona
  - One of a Kind Clinical Research Center LLC, Paradise Valley, Arizona
  - Mayo Clinic- Arizona, Scottsdale, Arizona
  - GI Alliance- Sun City, Sun City, Arizona
  - Adobe Clinical Research LLC, Tucson, Arizona
  - Gastroenterology and Liver Institute, Escondido, California
  - Om Research LLC, Lancaster, California
  - So. California Research Institute Med Group Inc./West Gastroenterology Med Group, Los Angeles, California
  - UCLA, Los Angeles, California
  - Providence Facey Medical Foundation, Mission Hills, California
  - Stanford University School of Medicine, Redwood City, California
  - Medical Associates Research Group, Inc., San Diego, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - Medical Research Center of Connecticut, LLC 300143562, Hamden, Connecticut
  - Central Connecticut Endoscopy Center, Plainville, Connecticut
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - University of Miami Medical Center, Miami, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - St. Johns Center for Clinical Research, Saint Augustine, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - Agile Clinical Research Trials, Alpharetta, Georgia
  - Lemah Creek Clinical Research, Oakbrook Terrace, Illinois
  - Indiana University -GI, Indianapolis, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical, Burlington, Massachusetts
  - Hawthorn Medical Associates LLC, South Dartmouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Revive Research Institute, Inc, Farmington Hills, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, School of Medicine, St Louis, Missouri
  - Manhattan Clinical Research, LLC, Manhattan, New York
  - New York University Medical Center PRIME, New York, New York
  - Blair S Lewis MD, New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Tryon Medical Partners, Charlotte, North Carolina
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Gastro Health Research, Cincinnati, Ohio
  - Cleveland Clinic - Gastroenterology and Hepatology, Cleveland, Ohio
  - Dayton Gastroenterology, Inc, Englewood, Ohio
  - Eastern Pennsylvania Gastroeneterology and Liver Specialists, Allentown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Rapid City Medical Center, LLC, Rapid City, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Methodist Hospital 150520246, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Spring Clinical Research, Houston, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Victoria Gastroenterology, Victoria, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Swedish Gastroenterology, Seattle, Washington
  - University of Washington Division of Gastroenterology, Seattle, Washington
  - Velocity Clinical Research, Spokane, Washington
- Belgium (3):
  - AZ Sint-Lucas, Bruges
  - AZ Maria Middelares, Ghent
  - Vitaz, Sint-Niklaas
- Canada (4):
  - Gastroenterology and Internal Medicine Research Institute (GIRI), Edmonton, Alberta
  - St. Boniface Hospital Inc. Section of Nephrology BG 007, Winnipeg, Manitoba
  - Kensington Screening Clinic, Toronto, Ontario
  - McGill University Health Center McGill University, Montreal, Quebec
- France (5):
  - Hopital Rangueil Service de Gastro Enterologie et Nutrition, Toulouse, Haute Garonne
  - Institut des MICI, Neuilly, Hauts De Seine
  - CHU Lille - Hopital Claude Huriez Service des maladies de I'appareil digestif, Lille, Nord
  - CHU Saint Etienne - Hopital Nord Service de Gastro-Enterologie et Hepatologie, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Hopital Europeen Georges Pompidou Gastro Enterologie et Oncologie Digestive, Paris
- Italy (10):
  - Azienda Ospedaliero Universitaria di Ferrara, Cona, Ferrara
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan, Milano
  - Azienda Ospedaliero Universitaria Ospedali Riuniti- Ospedale Pediatrico UOC Pediatria - G. Salesi, Ancona
  - Ospedale Valduce 300205849, Como
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Internal Medicine, Palermo
  - Fondazione IRCCS Policlinico San Matteo Sezione di Medicina Interna, Pavia
  - Azienda Ospedaliero Universitaria Pisana (Presidio di Cisanello) U.O. Gastroenterologia, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS UOC Medicina Interna e Gastroenterologia, Roma
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
  - Ospedale Umberto I di Torino S.C. Gastroenterologia, Torino
- Poland (8):
  - FutureMeds Krakow prev. Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - ALLMEDICA sp. z o. o., Nowy Targ
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Centrum Medyczne Medyk, Rzeszów
  - Warsaw IBD Point Profesor Kierkus, Warsaw
  - Komisja Bioetyczna przy Okregowej Izbie Lekarskiej w Warszawie, Warsaw
  - Melita Medical SP . Z O. O., Wroclaw
  - ETG Zamosc, Zamość
- Spain (5):
  - Vall d'Hebron Research Institute, Barcelona
  - Hospital Universitario Ramon y Cajal Servicio de Gastroenterologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria Digestive Service, Málaga
  - Hospital Universitario Virgen Macarena Digestive Service, Seville
  - Hospital Universitario Miguel Servet Servicio de Aparato Digestivo, Zaragoza
- United Kingdom (6):
  - Royal London Hospital Dept of Gastroenterology, London, Greater London
  - King's College Hospital Dept of Gastroenterology, London, Greater London
  - John Radcliffe Hospital Dept of Gastroenterology, Oxford, Oxfordshire
  - Royal Hallamshire Hospital Dept of Gastroenterology, Sheffield, South Yorkshire
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, West Yorkshire
  - The Ulster Hospital Department of Gastroenterology, Belfast

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click on this link — https://clinicaltrials.takeda.com/study-detail/44e4ec7deb684f49?idFilter=%5B%22TAK-062-2001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at various investigative sites globally from 30 June 2022 to 06 November 2024.
Pre-assignment Details: Participants with a diagnosis of celiac disease were enrolled and randomly assigned to receive either TAK-062 Placebo + simulated inadvertent gluten exposure (SIGE) Gluten-Bar or pre-determined amount of TAK-062 + SIGE Gluten-Bar in Cohort 1. 153 participants were enrolled in the trial but 1 participant out of 153 was randomized but not treated. Cohort 2 of the trial was not initiated.
Groups:
- Placebo + SIGE Gluten-Bar: Participants received TAK-062 placebo-matching tablets and SIGE gluten bar, orally for up to 24 weeks.
- TAK-062 + SIGE Gluten-Bar: Participants received pre-determined amount of TAK-062 tablets and SIGE gluten bar, orally, for up to 24 weeks.
Period: Overall Study
Arm/Group | Placebo + SIGE Gluten-Bar | TAK-062 + SIGE Gluten-Bar
Started | 76 | 77
Completed | 55 | 51
Not Completed | 21 | 26
Not completed — Adverse Event | 5 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 13 | 17
Not completed — Reason Not Specified | 1 | 0
Not completed — Randomized in Error & Not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS)- SIGE included all randomized participants who were randomized to receive gluten-containing SIGE.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + SIGE Gluten-Bar | TAK-062 + SIGE Gluten-Bar | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (15.35) | 46.8 (12.95) | 46 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 115
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 69 | 70 | 139
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 74 | 71 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Celiac Disease Symptom Diary (CDSD) Gastrointestinal (GI) Symptom Severity Score From Baseline to Week 12
Description: CDSD GI symptom severity score is an average of the daily GI symptom severity scores during the week. The daily GI symptom severity score is the average of the severity score for diarrhea, abdominal pain, bloating and nausea, ranging from 0 to 4. Symptom severity is evaluated using 5-point Likert-type scales (none, mild, moderate, severe, and very severe). Higher scores indicate more severe symptoms. Results are reported as least squares (LS) mean change from baseline at Week 12, determined using a mixed-effect model for repeated measures (MMRM). A negative change from baseline indicates improvement.
Time Frame: Baseline (Week -1) to Week 12
Population: The FAS-SIGE included all randomized participants who were randomized to receive gluten-containing SIGE. Overall number of participants analyzed is the number of participants with data available for analysis. Cohort 2 of the trial was not initiated.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + SIGE Gluten-Bar | TAK-062 + SIGE Gluten-Bar
Number analyzed (Participants) | 61 | 59
score on a scale | -0.128 (0.083) | -0.111 (0.082)
Statistical Analysis 1: Comparison: Placebo + SIGE Gluten-Bar vs TAK-062 + SIGE Gluten-Bar; Test type: Superiority; p = 0.847, MMRM — P-value was based on a MMRM analysis with treatment group, week, treatment-by-week interaction, & the randomization stratification factors as fixed effects & baseline CDSD GI symptom severity scores as covariates, and participant as a random effect; LS Mean Difference = 0.017, 95% CI 2-sided [-0.162 to 0.197]

2. Secondary Outcome: Change in Villous Height to Crypt Depth Ratio (Vh:Cd) From Baseline to Week 24
Description: The Vh:Cd ratio represents mucosal architectural changes and a lower Vh:Cd ratio indicates more severe intestinal injury characterized by a flattening of the mucosa. Results are reported as least squares (LS) mean change from baseline at Week 24, determined using an analysis of covariance (ANCOVA) model. A negative change from baseline indicates worsening disease.
Time Frame: Baseline (Week -4, Run-in Period) to Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: unitless ratio
Arm/Group | Placebo + SIGE Gluten-Bar | TAK-062 + SIGE Gluten-Bar
Number analyzed (Participants) | 60 | 59
unitless ratio | -0.006 (0.100) | -0.338 (0.099)
Statistical Analysis 1: Comparison: Placebo + SIGE Gluten-Bar vs TAK-062 + SIGE Gluten-Bar; Test type: Superiority; p < 0.001, ANCOVA — P-value was based on a ANCOVA model with treatment group and randomization stratification factors as fixed effects and baseline Vh:Cd as covariates; LS Mean Difference = -0.331, 95% CI 2-sided [-0.481 to -0.181]

3. Secondary Outcome: Percentage of Participants Experiencing at Least One Treatment-Emergent Adverse Event (TEAE), Serious Treatment-Emergent Adverse Events (Serious TEAEs) and Treatment-Related TEAEs
Description: Adverse event(AE)=any untoward medical occurrence in clinical investigation participant administered a drug; it does not necessarily have to have causal relationship with this treatment.AE can therefore be any unfavorable&unintended sign(e.g.,clinically significant abnormal laboratory value, electrocardiogram[ECG] value,or vital sign measurement),symptom,or disease temporally associated with use of drug whether or not it is considered related to drug.TEAE=new onset or worsening AEs after first dose of study treatment regardless of relationship to study drug.SAE=any untoward medical occurrence at any dose that results in death,is life threatening,requires inpatient hospitalization/prolongation of existing hospitalization,results in persistent/significant disability/incapacity,leads to a congenital anomaly/birth defect/is important medical event. TEAEs considered related to study drug as assessed by investigator were reported.Percentages were rounded off to nearest single decimal place.
Time Frame: Up to Week 28
Population: The Safety Analysis Set (SAF) included all randomized participants who received at least 1 dose of study drug. Cohort 2 of the trial was not initiated.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + SIGE Gluten-Bar | TAK-062 + SIGE Gluten-Bar
Number analyzed (Participants) | 76 | 76
percentage of participants
  TEAEs | 64.5 | 73.7
  Serious TEAEs | 5.3 | 1.3
  Treatment-Related TEAEs | 5.3 | 13.2

4. Secondary Outcome: Number of Participants With Positive Antidrug Antibodies (ADA) in Serum for TAK-062
Description: A positive ADA participant was defined as a participant who had at least 1 positive ADA result during the study and was further categorized as: Transiently positive- defined as participants with confirmed positive ADA in at least 1 sample and no consecutive samples; Persistently positive- defined as participants with confirmed positive ADA in 2 or more consecutive positive ADA samples.
Time Frame: Up to Week 28
Population: Immunogenicity Analysis Set included all randomized participants who received any TAK-062 and had the baseline and at least 1 postbaseline immunogenicity sample assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + SIGE Gluten-Bar | TAK-062 + SIGE Gluten-Bar
Number analyzed (Participants) | 76 | 76
Participants
  At least 1 Positive ADA | 27 | 67
  Transiently Positive | 19 | 8
  Persistently Positive | 8 | 59

ADVERSE EVENTS:
Time Frame: Up to Week 28
Description: The SAF included all randomized participants who received at least 1 dose of study drug.
Groups:
- TAK-062 Placebo + SIGE Gluten-Bar: Participants received TAK-062 placebo-matching tablets and SIGE gluten bar, orally for up to 24 weeks.
Arm/Group | TAK-062 Placebo + SIGE Gluten-Bar | TAK-062 + SIGE Gluten-Bar
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 4/76 | 1/76
Other Adverse Events (participants affected / at risk) | 13/76 | 24/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-062 Placebo + SIGE Gluten-Bar (N=76) | TAK-062 + SIGE Gluten-Bar (N=76)
ANASTOMOTIC COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-062 Placebo + SIGE Gluten-Bar (N=76) | TAK-062 + SIGE Gluten-Bar (N=76)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 5
DIARRHOEA (Gastrointestinal disorders) | 2 | 13
FATIGUE (General disorders) | 3 | 4
GASTRITIS (Gastrointestinal disorders) | 0 | 4
NAUSEA (Gastrointestinal disorders) | 3 | 4
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 2 | 4
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 4
VOMITING (Gastrointestinal disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT05353985/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT05353985/SAP_001.pdf